CLINICAL TRIAL: NCT01109251
Title: Post CVA Persistent Hypetension, Interest of Caring by Tensional Auto-measures
Brief Title: Post CVA Persistent Hypertension Caring
Acronym: Hippocrate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hippocrate
Record Dates: First submitted 2010-03-16; First posted 2010-04-23 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Post CVA Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Other): Group of patients presenting a non controlled AHT or a masked AHT, benefiting from an optimised caring at visit 0.
  Interventions: Procedure: Auto-measure of the tension by an autotensiometer
- Control group (Other): Patients presenting a non controlled AHT(persistent AHT, AHT necessiting an adaptation of the treatment by the generalist) with information of the generalist on the necessity of obtaining the tensional control according the HAS recommendations
  Interventions: Procedure: Auto-measure of the tension by an autotensiometer

INTERVENTIONS:
Procedure: Auto-measure of the tension by an autotensiometer — All hypertended patients able to realise a serie of tensional auto-measures will be invited to realise a serie of tensional auto-measures theree days before the consultation in the neurology department.
  The auto-measures will be performed according the methodology recommended by HAS.
  Arms: Intervention group
Procedure: Auto-measure of the tension by an autotensiometer — All hypertended patients able to realise a serie of tensional auto-measures will be invited to realise a serie of tensional auto-measures theree days before the consultation in the neurology department.
  The auto-measures will be performed according the methodology recommended by HAS.
  Arms: Control group

SUMMARY:
The study HIPPOCRATE is a prospective open comparative study with a control group.

The objective of this study is to show that an optimization of the caring of non controlled hypertended patients following a CVA (including a preliminary Tensional auto-measure (TAM) at the follow-up visit, an education of the patient with a decision support tree for the generalist and/or a visit in the multidisciplinary AHT department), allow to obtain a better tensional control copared to the usual caring.

DETAILED DESCRIPTION:
This study compares the usual follow up of patients seen at a visit three months following the CVA, with a optimised follow up including the tensional auto-measure, the education of the patient and the information of the generalist and the appeal to the AHT multidisciplinary visit for resistant patients, in compliance with the guidelines.

All the hypertended patients able to realise a course of tensional automeasures will be invited to realise a course of tensional auto-measures during three days preceding the visit in the neurology department.

The tensional measures will be performed according the methodology recommended by HAS.

This strategy of caring is conform to the HAS and ESH recommendations regarding the follow up of the hypertended patients.

The hospitalised patients in neurology for CVA are in all cases convocated to the follow up visit three months after the hospitalisation. The patients will be trained in the use of the TAM by the nurse of the neurology depratment before his dropout from the neurology department at the end of hospitalisation.

The systematic use of TAM will allow to identify patients presenting a AHT "white blouse", but too patients presenting masked AHT.

The visit in the neurology department will be performed by the investigators of the neurology department. At the end of this visit, two groups of patients will be identified : patients with a controlled AHT (NI), and patients with a masked or non controlled AHT (MASC + NC).

Patients presenting a controlled AHT or a "white blouse" AHT (NI) will not be randomised. But it will be proposed to them to sign a consent to acquire their agreement to realise a exploitation of their data. This will allow to caracterise better this population of patients.

Patients presenting a masked or non controlled AHT will be invited to participate to the study after signing a consent.

The collection of the consent will be done by the investigators of the neurology department.

ELIGIBILITY:
Inclusion Criteria:

Patient male or female from 20 to 80 years old included.

* ischemic or haemorragic CVA or TIA necessiting an hospitalisation or a consultation in the neurolgy department, from more than 2 months.
* Pression ≥140/90 ou 130/80 (diabetic) during the post CVA consultation and a mean TAM ≥135/85 ou 125/75 (diabetic) = non controlled AHT OR Pression < 140/90 ou 130/80 (diabetic) during the post CVA consultation and a mean TAM ≥ 135/85 ou 125/75 (diabetic) = masked AHT
* Patient agreed to participate to the study and having signed the informed consent from

Exclusion Criteria:

* malignant AHT necessiting the urgent and specialised caring
* Persistance of a carotids bilateral stenosis from more than 70%
* Severe Renal Insufficiency (Creatinin Clearance estimated by the formula MDRD < 30 ml/mn)
* CVA with major sequelae which according the judgement of the investigator will not allow to realise TAM :

  * Major Cognitive Troubles
  * Severe motor Troubles
* Severe concomitant Pathology
* Patient not speaking and not understanding french.
* Contre-indications to the realisation of TAM :

  * Cardiac Arythmy
  * Obese Patients for which the circumference of the arm is > 33 cm
* Patient refusing to go to the 3 months after hospitalisation follow up consultation.
* Patient with no identified generalist
* Patient refusing to sign the informed consent form.
* Absence of affiliation to a Social system.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
tensional auto-measure | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nancy, Nancy, France
  - CH Bar Le Duc, Bar-le-Duc